CLINICAL TRIAL: NCT07014761
Title: The Influence of Central Sensitization in Endometriosis Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2025-195-02
Record Dates: First submitted 2025-04-26; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis; Adenomatosis
Keywords: central sensitization;; endometriosis;; adenomyosis
MeSH Terms: conditions — Endometriosis; Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CS group: CS group（CSI score ≥40 ）
  Interventions: Other: No Intervention: Observational Cohort
- no CS group: no CS group (CSI score <40).
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention

SUMMARY:
Endometriosis diseases include endometriosis and adenomyosis. Researchers will include 200 or more patients with endometriosis diseases; collect relevant clinical data such as age, BMI, educational level, history of other diseases, surgical history, smoking and drinking history, pregnancy and childbirth history, pain duration, preoperative CA125 level, hemoglobin, surgical methods (laparotomy / laparoscopy), endometriosis stage, endometriosis location, baseline (preoperative), 1, 3, and 6-month follow-up CSI scores, dysmenorrhea scores, chronic pelvic pain scores, dyspareunia scores, dyschezia scores, back pain scores, to explore the role of central sensitization in postoperative pain of patients with adenomyosis, that is, the relationship between central sensitization and postoperative pain outcomes (chronic pelvic pain, dyspareunia, dyschezia, back pain); evaluate whether the baseline CSI score can predict the severity of postoperative pain; and explore the pain relief of different medications after lesion resection in patients with endometriosis.

DETAILED DESCRIPTION:
Endometriosis and adenomyosis are included in endometriotic diseases. Endometrial tissue appears outside the uterine is called endometriosis. Adenomyosis is a common gynecological disease in reproductive-aged women. Its characteristic is that endometrial glands and stroma invade the uterine myometrium, accompanied by the proliferation of surrounding smooth muscle cells. 20.9% to 34% of reproductive-aged women have adenomyosis detected by ultrasound examination. Most patients with endometriotic diseases will experience various forms of pain, such as dysmenorrhea, dyspareunia, chronic pelvic pain (CPP) , dyschezia, or back pain, etc. Surgical treatment (such as lesion resection, hysterectomy) is still a common method for treating endometriotic diseases. However, some patients still have persistent pain after surgery.

The mechanism of central sensitization (CS) may explain why about 30% of endometriosis patients have persistent CPP after traditional surgical treatment. Previous study indicates that almost half of endometriosis patients (42%) have CS, and CS is independently associated with moderate to severe chronic pelvic pain, and the score of the Central Sensitization Inventory (CSI) at the baseline before surgery is significantly correlated with persistent CPP after surgery. Therefore, it is reasonable to speculate that central sensitization may also be a potential cause of persistent pain after adenomyosis surgery. However, there is currently no relevant study indicating whether central sensitization plays a role in persistent pain after hysterectomy in adenomyosis patients, nor is there any relevant study indicating the pain relief of different medications after lesion resection in endometriosis patients. In this study, researchers will include 200 or more patients with endometriosis diseases; collect relevant clinical data such as age, BMI, educational level, history of other diseases, surgical history, smoking and drinking history, pregnancy and childbirth history, pain duration, preoperative CA125 level, hemoglobin, surgical methods (laparotomy / laparoscopy), endometriosis stage, endometriosis location, baseline (preoperative), 1, 3, and 6-month follow-up CSI scores, dysmenorrhea scores, CPP scores, dyspareunia scores, dyschezia scores, back pain scores. By applying appropriate statistical methods, such as the Mann-Whitney U test or Kruskal-Wallis test for continuous variables, and the Pearson χ2 test for categorical variables, researchers will explore the role of central sensitization in pain after hysterectomy in adenomyosis patients, explore the pain relief of different medications after lesion resection in endometriosis patients, and provide new ideas for postoperative pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the gynaecological ward of Sun Yat-sen Memorial Hospital from March 2025 to March 2027;
2. Age 18-50 years old;
3. Endometriosis focus excision or hysterectomy (with or without bilateral salpingo-oophorectomy, with excision of any complicated lesion);
4. The pathology was adenomyosis or endometriosis.

Exclusion Criteria:

1. Postmenopausal (spontaneous or surgical);
2. Hysterectomy and/or bilateral salpingo-oophorectomy (before baseline)
3. Lack of CSI or CPP score;
4. The postoperative follow-up time was less than 6 months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will include 200 or more patients with endometriosis diseases; these patients are admitted to the gynaecological ward of Sun Yat-sen Memorial Hospital from March 2025 to March 2027; aged 18-50 years old; endometriosis focus excision or hysterectomy (with or without bilateral salpingo-oophorectomy, with excision of any complicated lesion); the pathology was adenomyosis or endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
central sensitization inventory score | pre-operation；1, 3, 6 months after surgery
  The central sensitization inventory score (0 to 100) was obtained by central sensitization inventory questionnaire; a higher score indicates greater symptom severity that may be indirectly related to conditions with underlying central sensitization

SECONDARY OUTCOMES:
dysmenorrhea scores | pre-operation；1, 3, 6 months after surgery
  the pain scores were rated on an 11-point numeric rating scale (0-10, with 0 indicating no pain and 10 indicating worst pain imaginable)
chronic pelvic pain scores | pre-operation；1, 3, 6 months after surgery
  the pain scores were rated on an 11-point numeric rating scale (0-10, with 0 indicating no pain and 10 indicating worst pain imaginable)
dyspareunia scores | pre-operation；1, 3, 6 months after surgery
  the pain scores were rated on an 11-point numeric rating scale (0-10, with 0 indicating no pain and 10 indicating worst pain imaginable)
dyschezia scores | pre-operation；1, 3, 6 months after surgery
  the pain scores were rated on an 11-point numeric rating scale (0-10, with 0 indicating no pain and 10 indicating worst pain imaginable)
back pain scores | pre-operation；1, 3, 6 months after surgery
  the pain scores were rated on an 11-point numeric rating scale (0-10, with 0 indicating no pain and 10 indicating worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Yingchen Wu, Doctor, Study Director — 中山大学孙逸仙纪念医院
Locations (1):
- Sun Yat-sen Memorial Hospital，Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
No URL available at this time

REFERENCES:
- [Background] Harada T, Taniguchi F, Guo SW, Choi YM, Biberoglu KO, Tsai SS, Alborzi S, Al-Jefout M, Chalermchokcharoenkit A, Sison-Aguilar AG, Fong YF, Senanayake H, Popov A, Hestiantoro A, Kaufman Y. The Asian Society of Endometriosis and Adenomyosis guidelines for managing adenomyosis. Reprod Med Biol. 2023 Sep 10;22(1):e12535. doi: 10.1002/rmb2.12535. eCollection 2023 Jan-Dec. PMID 37701076
- [Background] Raimondo D, Raffone A, Renzulli F, Sanna G, Raspollini A, Bertoldo L, Maletta M, Lenzi J, Rovero G, Travaglino A, Mollo A, Seracchioli R, Casadio P. Prevalence and Risk Factors of Central Sensitization in Women with Endometriosis. J Minim Invasive Gynecol. 2023 Jan;30(1):73-80.e1. doi: 10.1016/j.jmig.2022.10.007. Epub 2022 Oct 29. PMID 36441085
- [Background] Orr NL, Huang AJ, Liu YD, Noga H, Bedaiwy MA, Williams C, Allaire C, Yong PJ. Association of Central Sensitization Inventory Scores With Pain Outcomes After Endometriosis Surgery. JAMA Netw Open. 2023 Feb 1;6(2):e230780. doi: 10.1001/jamanetworkopen.2023.0780. PMID 36848090
- [Background] Orr NL, Wahl KJ, Lisonek M, Joannou A, Noga H, Albert A, Bedaiwy MA, Williams C, Allaire C, Yong PJ. Central sensitization inventory in endometriosis. Pain. 2022 Feb 1;163(2):e234-e245. doi: 10.1097/j.pain.0000000000002351. PMID 34030173

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT07014761/Prot_SAP_000.pdf